CLINICAL TRIAL: NCT05008237
Title: Weekly Docetaxel Plus Cisplatin as First-line Chemotherapy in Metastatic Salivary Gland Cancer Patients : a Multicenter Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-07-149
Record Dates: First submitted 2021-01-13; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Salivary Gland Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cisplatin plus docetaxel (Experimental): D1, D8 Docetaxel 35 mg/m2 + D5W 100mL MIV over 1hr D1 Cisplatin 70mg/m2 + NS 150mL MIV over 1hr every 3 weeks
  Treatment will be continued until disease progression or unacceptable toxic effects.
  Interventions: Drug: docetaxel plus Cisplatin

INTERVENTIONS:
Drug: docetaxel plus Cisplatin — D1, D8 Docetaxel 35 mg/m2 + D5W 100mL MIV over 1hr D1 Cisplatin 70mg/m2 + NS 150mL MIV over 1hr every 3 weeks Treatment will be continued until disease progression or unacceptable toxic effects.

SUMMARY:
Cisplatin plus weekly docetaxel as first-line chemotherapy in metastatic salivary gland cancer patients : a multicenter phase II study

DETAILED DESCRIPTION:
Preclinically, paclitaxel and docetaxel have demonstrated activity against salivary gland cancers1. Phase II trial of single-agent paclitaxel2, conducted by Eastern Cooperative Oncology Group in 45 patients with advanced SGC. Eight partial responses were observed among the 31 patients with mucoepidermoid carcinoma (MEC) or adenocarcinoma, but no responses were identified in the 14 patients with ACC. Based on its impressive anti-tumor activity in patients with head and neck cancer, especially in squamous cell carcinoma, Ragusa et al.3 evaluated the activity of docetaxel in 4 patients with high grade MEC of the major salivary glands. The treatment was well tolerated, and there was complete response in two and partial response in the other two patients.

However, myelosuppression is one of the serious concerns with every 3 week schedule of docetaxel administration, especially in older patients. Alternatively, a weekly dosing of docetaxel has been reported to reduce toxicity and Investigator previously reported weekly docetaxel and cisplatin chemotherapy in recurrent or metastatic nasopharyngeal cancer demonstrated high response rate with modest toxicities4. So Investigator planned this phase II study to evaluate the efficacy and safety of cisplatin plus weekly docetaxel in patients with metastatic salivary gland cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed salivary gland cancer with one of the following histologic subtypes : mucoepidermoid, adenocarcinoma/ductal carcinoma or adenoid cystic carcinoma

  * Only progressive disease in case of ACC

    * Progressive disease is defined as one of the following occurring within 6 months of study entry (i) at least a 20% increase in radiologically or clinically measurable disease, (ii) appearance of new lesions or (iii) deterioration in clinical status

      * stage IV or recurrent cancer which is incurable with surgery or radiotherapy

        * age ≥ 20 years

          * ECOG performance status 0-1 ⑥ At least one measurable tumor lesion according to RECIST 1.1

            * Expected survival for approximately 12 weeks or longer

              ⑧ No prior systemic chemotherapy (Patients who received adjuvant chemotherapy or chemoradiotherapy completed more than 6 months before will be eligible)
              * At least 4 weeks later after major surgery or radiotherapy ⑩ Organ function as evidence by the following; WBC ≥ 3,500 cells/mm3 and ≤ 50,000 cells/mm3, ANC ≥ 1,500 cells/mm3, Hemoglobin ≥ 10 g/dL (transfusion allowed), Platelet count ≥ 100,000 plts/mm3; Total bilirubin ≤ 1.5 ULN AST/ALT ≤ 2.5 ULN, (if liver metastases: AST, ALT ≤5.0 x ULN); Creatinine clearance 50 mL/min or serum creatinine ≤ 1.5 x UNL ⑪ Written informed consent

Exclusion Criteria:

* Severe or unstable cardiac disease, including (for example) coronary artery disease requiring increased doses of anti-anginal medication and/or coronary angioplasty (including stent placement) within the preceding 24 months (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction within the last twelve months, significant arrhythmias)

  * Uncontrolled systemic illness such as DM, hypertension, hypothyroidism and infection

    * Pregnant and nursing women (women of reproductive potential have to agree to use an effective contraceptive method) ④ Symptomatic CNS malignancy (history of completely resected or irradiated brain metastases by WBRT or stereotactic radiosurgery allowed) ⑤ Patients with alcohol abuse

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05-02 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Response rate | Up to 30months
  To evaluate the effectiveness of regimen. The overall response rate will be measured by RECIST v1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | The time until defineded by date of all-cause mortality from date of IP administration. Up to 30 months.
  Overal survival defined by date of all-cause mortality from date of IP administration will be calculated.
progression-free survival (PFS) | The time until the date of either disease progression or the all cause mortality from the date of IP administration. Up to 30months.
  It is measure of the period of survival without disease progression.
Adeverse event(AE) | from the date of informed consent signature to 21days after last drug administration.
  Adverse event will be evaluate using CTCAE V.4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnamgu, South Korea